CLINICAL TRIAL: NCT03896646
Title: Radioembolization for HCC Patients With Personalized Yttrium-90 Dosimetry for Curative Intent (RAPY90D)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1008; NCI-2019-01586 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1008 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Stage III Hepatocellular Carcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (personalized radioembolization, SPECT/CT HIDA) (Experimental): Patients undergo yttrium-90 microsphere radioembolization with yttrium Y 90 glass microspheres using personalized dose measurements. Patients also undergo SPECT/CT HIDA scan before radioembolization and 2-4 months after radioembolization.
  Interventions: Procedure: Computed Tomography; Other: Hepatobiliary Iminodiacetic Acid Scan; Procedure: Single Photon Emission Computed Tomography; Radiation: Yttrium Y 90 Glass Microspheres; Procedure: Yttrium-90 Microsphere Radioembolization

INTERVENTIONS:
Procedure: Computed Tomography — Undergo SPECT/CT HIDA scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Other: Hepatobiliary Iminodiacetic Acid Scan — Undergo SPECT/CT HIDA scan
  Other Names: HIDA Scan
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT HIDA scan
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Radiation: Yttrium Y 90 Glass Microspheres — Undergo radioembolization with yttrium Y 90 glass microspheres
  Other Names: TheraSphere
Procedure: Yttrium-90 Microsphere Radioembolization — Undergo yttrium-90 microsphere radioembolization
  Other Names: Yttrium Y 90 Microsphere Therapy; Yttrium-90 Radioembolization

SUMMARY:
This trial aims to improve hepatocellular carcinoma (HCC) tumor responses in patients undergoing Y90 radioembolization by using personalized dosimetry as part of treatment planning. Using standard calculations for Y90 doses may not be specific enough for individual patients given that there can be differences in how tumor cells and liver cells respond to radiation. Personalized dose plans may help improve treatment and outcomes in liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To achieve tumor objective response rates of 75% using voxel based dosimetry when the mean dose (Dmean) to tumor is targeted to be greater than 200 Gray (Gy).

SECONDARY OBJECTIVES:

I. Correlate changes in liver function and Common Terminology Criteria for Adverse Events (CTCAE) incidence to the mean absorbed dose to normal liver.

II. Prospectively validate the accuracy of our published tumor dose response prediction based on the yttrium Y 90 glass microspheres (yttrium-90 [Y90]) tumor dose volume histograms (DVHs).

III. Correlate predicted tumor doses macroaggregated albumin (MAA) scan with actual doses delivered (Y90 scan).

IV. Develop a tumor dose response model prediction based on the MAA dose maps. V. Develop a model correlating normal liver radiation dose to liver function using single-photon emission computed tomography/computed tomography hepatobiliary iminodiacetic acid (SPECT/CT HIDA) imaging.

VI. Develop a model correlating the relative tumor to normal liver enhancement on CT imaging and Cone beam CT imaging to the uptake on SPECT CT Tc99m MAA imaging (gold standard).

VII. Compare tumor and normal liver doses estimations from SPECT CT Bremsstrahlung imaging to positron emission tomography (PET) CT imaging.

OUTLINE:

Patients undergo yttrium-90 microsphere radioembolization with yttrium Y 90 glass microspheres using personalized dose measurements. Patients also undergo SPECT/CT HIDA scan before radioembolization and 2-4 months after radioembolization.

After completion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age, of any race or sex, who have unresectable hepatocellular carcinoma of the liver, and who are able or have a fully able legal guardian to give informed consent, will be eligible. Patients must have an ECOG Performance Status score of </=2, with a life expectancy of >/=3 months, and must be non-pregnant with an acceptable contraception in premenopausal women. Patients must be >4 weeks since prior radiation or prior surgery and at least one month post chemotherapy.
2. At least one lesion >/= 3.0 cm in shortest dimension
3. AST or ALT <5 times ULN
4. Bilirubin </= 2.0 mg/dL (unless segmental infusion is used)
5. Negative pregnancy test in premenopausal women

Exclusion Criteria:

1. Contraindications to angiography and selective visceral catheterization
2. Evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) to the lungs with a single injection, or greater than 50 Gy for multiple injections
3. Evidence of any detectable Tc-99m MAA flow to the stomach or duodenum, after application of established angiographic techniques to stop or mitigate such flow (eg, placing catheter distal to gastric vessels)
4. Significant extrahepatic disease representing an imminent life-threatening outcome
5. Severe liver dysfunction or pulmonary insufficiency
6. Active uncontrolled infection
7. Significant underlying medical or psychiatric illness
8. Pregnant
9. Pre-existing diarrhea/illness, co-morbid disease or condition that would preclude safe delivery of TheraSphere® treatment and place the patient at undue risk
10. Infiltrative tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Tumor objective response rate (ORR) | Up to 6 months
  Assessed with modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria. The ORR of treated tumors will be determined. Will perform a cluster bootstrap in which patients (not tumors) are sampled with replacement. Will construct a 95% confidence interval using the 2.5% and 97.5% quantiles of the bootstrap sampling distribution.

SECONDARY OUTCOMES:
Changes in liver function | Up to 6 months
  Will analyze the correlation in changes in liver function to the mean absorbed dose to normal liver. The hepatobiliary iminodiacetic acid (HIDA) scan will be used to estimate the body-surface area corrected mebrofenin clearance rate in %-activity/sec/m^2 using published methodology. The change in liver function after radioembolization will be calculated and correlated to the radiation dose distribution to the normal liver. Will use Wilcoxon and two-sample t-tests to measure significance of association.
Changes in Common Terminology Criteria for Adverse Events (CTCAE) incidence | Up to 6 months
  Will analyze the correlation in changes in CTCAE incidence to the mean absorbed dose to normal liver. Will create waterfall charts of CTCAE and mean absorbed normal liver in liver. Will use Wilcoxon and two-sample t-tests to measure significance of association and scatterplots and regression (linear or non-linear) to predict actual doses delivered from predicted tumor dose.
Accuracy of published tumor dose response prediction based on the yttrium-90 (Y90) tumor dose volume histograms | Up to 6 months
  Lin's concordance correlation, t-test, and Bland-Altman analysis will be performed on pair-wise estimate of tumor doses. Develop tumor dose response curves using logistic regression and assess significance of parameters. Furthermore, we will compute the half-maximal dose (D50%), positive predictive value, negative predictive value and its 95% confidence interval from this prospective study. These values will be compared to those from the retrospective study for equivalence using the z-test.
Prediction of tumor doses macroaggregated albumin (MAA) scan with actual doses delivered (Y90 scan) | Up to 6 months
  Lin's concordance correlation, t-test, and Bland-Altman analysis will be performed on pair-wise estimate of tumor doses. Will use scatterplots and regression (linear or non-linear) to predict actual doses delivered from predicted tumor dose. A correlation analysis of the predicted tumor doses from the MAA images with the actual tumor doses delivered from Y90 images will be performed. The linear-correlation coefficient will be computed. A Bland-Altman analysis will be performed to compute the bias and the 95% limits of agreement.
Development of tumor dose response model prediction based on MAA dose maps | Up to 6 months
  Mean tumor doses based the planning 99mTc-MAA images will be computed using voxel dosimetry. A univariate logistic regression model will used to determine tumor dose metrics (D50%) that correlated with mRECIST-based tumor response at 3 and 6 months.
Development of a model correlating normal liver radiation dose to liver function using single-photon emission computed tomography computed tomography hepatobiliary iminodiacetic acid (SPECT CT HIDA) imaging | Up to 6 months
  A regression analysis of the change in liver function from the pre- and post-procedural HIDA SPECT/CT scans (changes in %/min) as a function of the normal liver absorbed dose will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Armeen Mahvash, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org